CLINICAL TRIAL: NCT00684723
Title: A Single Dose Crossover Comparative Bioavailability Study of Lovastatin 40mg Tablets in Healthy Male Volunteers/Fed State
Brief Title: Fed Bioavailability Study of Lovastatin Tablets and Mevacor Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Kristin Arnold, Vice President R&D, Mutual Pharmaceutical
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: LVI-P4-126
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Results first posted 2009-12-30 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Therapeutic Equivalency
MeSH Terms: interventions — Lovastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lovastatin 40 mg Tablet (Experimental): A single dose of Lovastatin 40 mg administered under fed conditions.
  Interventions: Drug: Lovastatin 40 mg Tablets
- Lovastatin (Mevacor®) 40 mg Tablet (Experimental): A single dose of Lovastatin (Mevacor®) 40 mg administered under fed conditions.
  Interventions: Drug: Lovastatin (Mevacor®) 40 mg Tablets

INTERVENTIONS:
Drug: Lovastatin 40 mg Tablets — 40 mg tablet administered 30 minutes following the start of a standardized high-fat, high-calorie breakfast
  Arms: Lovastatin 40 mg Tablet
Drug: Lovastatin (Mevacor®) 40 mg Tablets — 40 mg tablet administered 30 minutes following the start of a standardized high-fat, high-calorie breakfast
  Other Names: Mevacor®
  Arms: Lovastatin (Mevacor®) 40 mg Tablet

SUMMARY:
The purpose of this study is to evaluate and compare the relative bioavailability and therefore the bioequivalence of a test formulation of Lovastatin tablets to an equivalent dose of Mevacor® tablets after a single oral dose administered under fed conditions.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the relative bioavailability and therefore the bioequivalence of a test formulation of Lovastatin tablets to an equivalent dose of Mevacor® tablets after a single oral dose administered under fed conditions.

Fifty-four healthy, light/non/or ex-smoking, non-obese, male volunteers at least 18 years of age will be randomly assigned in a crossover fashion to receive each of two Lovastatin dosing regimens in sequence with a 7 day washout period between dosing periods. On the morning of Day 1, after an overnight fast of at least 10 hours, subjects will receive a standardized high-fat, high-calorie meal 30 minutes before drug administration. Thirty minutes after the start of the breakfast, a single oral dose of either the test formulation, Lovastatin (1 x 40 mg tablet), or a single oral dose of the reference formulation, Mevacor® (1 x 40 mg tablet) will be administered. After a 7 day washout period, on the morning of Day 8, following an overnight fast of at least 10 hours and 30 minutes after the start of a standardized high-fat, high-calorie meal, subjects will receive the alternate regimen. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of Lovastatin. Blood sampling will then continue on a non-confined basis at 36 and 48 hours post-dose. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout the confinement portion of the study for adverse reactions to the study drug and/or procedures. Vital signs will be monitored if judged necessary by the physician in charge. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Availability of volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form (ICF) duly signed by the volunteer
* Male aged of at least 18 with a body mass index (BMI) greater than or equal to 19 and below 30 kg/m²
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance
* Healthy according to the laboratory results and physical examination
* Light-, non- or ex-smokers. Light smokers are defined as someone smoking 10 cigarettes or less per day, and ex-smokers are defined as someone who completely stopped smoking for at least 3 months
* The informed consent must be signed by all volunteers, prior to their participation in the study

Exclusion Criteria:

* Significant history of hypersensitivity to lovastatin or any related products as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability, including but not limited to cholecystectomy
* Presence of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease
* Presence of active liver disease or unexplained persistent elevations of serum transaminases
* Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (>3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any clinically significant illness in the previous 28 days before day 1 of this study
* Use of enzyme-modifying drugs in the previous 28 days before day 1 of this study (all barbiturates, corticosteroids, phenylhydantoins, etc.)
* Participation in another clinical trial in the previous 28 days before day 1 of this study
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study
* Positive urine screening of drugs of abuse
* Positive results to HIV, HBsAg or anti-HCV tests

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-07; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma, Montreal, Quebec, Canada

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Lovastatin 40 mg Tablets Then Mevacor® 40 mg Tablets: On the morning of Day 1, subjects received one tablet of the test formulation, Lovastatin 40 mg, thirty minutes after the start of a standardized high-fat, high-calorie breakfast. After a 7 day washout period, on the morning of Day 8, subjects received one tablet of the reference formulation, Mevacor® 40 mg, thirty minutes after the start of a standardized high-fat, high-calorie breakfast.
- Mevacor® 40 mg Tablets Then Lovastatin 40 mg Tablets: On the morning of Day 1, subjects received one tablet of the reference formulation, Mevacor® 40 mg, thirty minutes after the start of a standardized high-fat, high-calorie breakfast. After a 7 day washout period, on the morning of Day 8, subjects received one tablet of the test formulation, Lovastatin 40 mg, thirty minutes after the start of a standardized high-fat, high-calorie breakfast.
Period: First Intervention
Arm/Group | Lovastatin 40 mg Tablets Then Mevacor® 40 mg Tablets | Mevacor® 40 mg Tablets Then Lovastatin 40 mg Tablets
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Lovastatin 40 mg Tablets Then Mevacor® 40 mg Tablets | Mevacor® 40 mg Tablets Then Lovastatin 40 mg Tablets
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Lovastatin 40 mg Tablets Then Mevacor® 40 mg Tablets | Mevacor® 40 mg Tablets Then Lovastatin 40 mg Tablets
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lovastatin 40 mg Tablets and Mevacor® 40 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either Lovastatin 40 mg or Mevacor® 40 mg thirty minutes after the start of a standardized high-fat, high-calorie breakfast.
Arm/Group | Lovastatin 40 mg Tablets and Mevacor® 40 mg Tablets
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.5, 5, 5.5, 6, 7, 8, 10, 14, 18, 24, 36, and 48 hours after drug administration.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Lovastatin 40 mg Tablets; Mevacor® 40 mg Tablets: On the morning of Day 1, subjects received one tablet of either the test formulation, Lovastatin 40 mg, or the reference formulation, Mevacor® 40 mg, thirty minutes after the start of a standardized high-fat, high-calorie breakfast. After a 7 day washout period, on the morning of Day 8, subjects received the alternate regimen thirty minutes after the start of a standardized high-fat, high-calorie breakfast.
Arm/Group | Lovastatin 40 mg Tablets | Mevacor® 40 mg Tablets
Number analyzed (Participants) | 54 | 54
ng/mL | 9.26 (6.13) | 10.01 (7.06)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Lovastatin 40 mg Tablets | Mevacor® 40 mg Tablets
Number analyzed (Participants) | 54 | 54
ng-hr/mL | 47.86 (29.34) | 51.64 (33.05)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Lovastatin 40 mg Tablets | Mevacor® 40 mg Tablets
Number analyzed (Participants) | 54 | 54
ng-hr/mL | 48.72 (29.14) | 52.98 (34.38)

ADVERSE EVENTS:
Groups:
- Lovastatin 40 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either Lovastatin 40 mg or Mevacor® 40 mg thirty minutes after the start of a standardized high-fat, high-calorie breakfast.
- Mevacor® 40 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either Lovastatin 40 mg or Mevacor® 40 mg thirty minutes after the start of a standardized high-fat, high- calorie breakfast.
Arm/Group | Lovastatin 40 mg Tablets | Mevacor® 40 mg Tablets
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 25/54 | 20/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovastatin 40 mg Tablets (N=54) | Mevacor® 40 mg Tablets (N=54)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry throat (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site edema (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0)
Edema peripheral (General disorders) | 1 (1) | 0 (0)
Venipuncture site bruise (General disorders) | 2 (2) | 0 (0)
Venipuncture site swelling (General disorders) | 1 (1) | 1 (1)
Burn esophageal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 2 (2)
Eosinophil count increased (Investigations) | 3 (3) | 3 (3)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Neutrophil count increased (Investigations) | 3 (3) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Somnolence (Nervous system disorders) | 9 (9) | 5 (5)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Vascular disorders) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days